CLINICAL TRIAL: NCT07050472
Title: Durvalumab as Consolidation Therapy After Concurrent Chemoradiotherapy (cCRT) for Patients With Limited-stage Small-cell Lung Cancer (LS-SCLC): A Retrospective, Single-center, Real-world Cohort Study
Brief Title: Durvalumab After Concurrent Chemoradiotherapy (cCRT) for Limited-stage Small-cell Lung Cancer (LS-SCLC)
Status: Completed | Type: Observational
Sponsor: Anhui Shi, MD (Other)
Responsible Party: Sponsor-Investigator, Anhui Shi, MD, chief physician, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Other Study IDs: 2025YJZ41
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Small-cell Lung Cancer
Keywords: limited stage small-cell lung cancer; CRT; immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- LS-SCLC

SUMMARY:
This is a retrospective, single-center study evaluating the effectiveness and safety of consolidative durvalumab after cCRT in LS-SCLC in real-world setting.

DETAILED DESCRIPTION:
Eligible LS-SCLC patients who received cCRT, and subsequent durvalumab from January 1st, 2020 till December 31st, 2023 will be identified and included for retrospective data collection and analyses in this study. Approximately 35~45 patients are planned to be enrolled. The first date of the presence of durvalumab treatment will be considered the index date for patients. Data is planned to be collected from date of histologically diagnosis up to June 27, 2025. The primary endpoint real-world PFS is defined as the time from the index date to disease progression (determined based on either radiological or clinical evidence) or death for any reason. Duration of durvalumab treatment and 2 year (relative to the first dose of durvalumab) rwPFS rate and OS rate will be measured.

Study data will come from what have been generated from routine clinical practice in the study hospital, e.g., the diagnosis, treatment and tumor assessments (CT or MRI, usually every 3 months for years 1~2, and every 6 months for years 3~5) information. Data collection, cleaning, and query will follow the traditional clinical study execution process. Investigators at study site will be responsible to ensure that data is accurate, clear, and traceable.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 at initial diagnosis.
2. Histologically or cytologically documented limited-stage SCLC (Stage I-III SCLC [T any, N any, M0] according to the American Joint Committee on Cancer Staging Manual [AJCC Cancer Staging Manual, 9th Edition] or the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology [IASLC Staging Manual in Thoracic Oncology 2016]).
3. Received concurrent chemoradiotherapy (cCRT) as first-line treatment and consolidative durvalumab prior to disease progression or death:

   * Received 4 cycles of platinum-based chemotherapy concurrent with radiotherapy.
   * The chemotherapy regimen must contain carboplatin/cisplatin and etoposide.
   * Received a total dose of radiation of 60 to 66 Gy over 6 weeks for standard QD radiation schedules, 45 Gy over 3 weeks or a simultaneous integrated boost of 54 Gy over 3 weeks for hyperfractionated BID radiation schedules.
   * Radiotherapy must have commenced no later than the end of Cycle 2 of chemotherapy.
   * Received at least 1 dose of durvalumab. The first dose of durvalumab received between 1 Jan 2020 and 31 Dec 2023 at Peking University Cancer Hospital.

Exclusion Criteria:

1. Mixed SCLC and NSCLC histology.
2. Participated in other interventional clinical trial for the treatment of any cancer during durvalumab therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically documented limited-stage SCLC (Stage I-III SCLC [T any, N any, M0] according to the American Joint Committee on Cancer Staging Manual [AJCC Cancer Staging Manual, 9th Edition] or the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology [IASLC Staging Manual in Thoracic Oncology 2016]).
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
rwPFS | Up to 60 months
  From the start of Durvalumab treatment to disease progression (tumor assessed by investigator) or death for any reason

SECONDARY OUTCOMES:
DoT | Up to 60 months
  Time from the start of Durvalumab treatment to the date of durvalumab discontinuation or death
real-world progression free survival rate at 24 months(rwPFS24) | 24 months after first dose of durvalumab
  Kaplan-Meier estimate of rwPFS (assessed by investigator) at 24 months after first dose of durvalumab
overall survival rate at 24 months (OS24) | 24 months after first dose of durvalumab
  Kaplan-Meier estimate of OS (assessed by investigator) at 24 months after first dose of durvalumab

OTHER OUTCOMES:
Adverse Events | From the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment
  AEs that occurred from the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China